CLINICAL TRIAL: NCT04920162
Title: Search for New Predictive Markers of the Immune Response in Vitiligo and Melanoma (Vitilimel Study)
Brief Title: Search for New Predictive Markers of the Immune Response in Vitiligo and Melanoma
Acronym: VITILIMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-AOIP-03
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Melanoma and Vitiligo
MeSH Terms: conditions — Melanoma; Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin deseases biospecimens collection (Other): Collect of blood samples without DNA into patients who had a vitiligo or a melanoma at day 0 until 1 year after their treatment
  Interventions: Other: Biospecimen into patients who had skin diseases

INTERVENTIONS:
Other: Biospecimen into patients who had skin diseases — Collect of blood samples without DNA into patients who had a vitiligo or a melanoma at day 0 until 1 year after their treatment

SUMMARY:
Skin diseases can have various origins. However, a number of them are linked to an imbalance in the immune system which will lead to either an excessively strong autoimmune response or a complete lack of response against cancer cells. Indeed, both melanoma and vitiligo are pathologies where the immune system plays an important role in the progression of the disease.

Advanced stage melanoma (metastatic lymph node and / or visceral) have a poor prognosis. Although targeted therapies and immunotherapies have improved the outcome for patient however significant proportion of these patients (~ 50%) developed resistance to therapies.

Vitiligo is a relatively common dermatosis affecting approximately 0.5% to 1% of the French population. Vitiligo results from the destruction of the melanocytes by the immune system. It is manifested by acquired depigmented macules, well limited and asymptomatic. Patients suffering from this condition have a marked decrease in their quality of life. There has been shown a strong link between vitiligo and melanoma. Indeed, patients with melanoma who develop vitiligo (~ 9% of patients treated with anti-PD-1 drugs) have a better prognosis compared to patients who do not develop vitiligo.

Interestingly, in melanoma cases where the immune system is inactive, the investigators have identified a new molecule secreted by melanoma cells, ITGBL1, leading to the exclusion of immune cells, decreased cytokines secretion and decreased immune cell activation. It is therefore essential to better understand the regulatory mechanism of the immune system in patients with vitiligo or in patients with melanoma treated by immunotherapy in order to be able to propose new therapeutic solutions for these patients.

No study to date has investigated the expression of ITGBL1 and serum inflammatory markers during the development of melanoma. Likewise in vitiligo, if a loss of ITGBL1 is observed, new treatments could be developed in order to limit the progression of the disease by re-expressing this protein.

Thus, the investigators exploratory study will provide the first answers to the predictive value of these markers for these pathologies in order to adapt and develop new treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with non-segmental vitiligo (vitiligo)
* Vitiligo affecting more than 5% of the total body surface (vitiligo)
* Patient with unresectable stage III or stage IV skin melanoma confirmed histologically (melanoma)
* Treatment-naïve patient with an indication for anti-PD1 mono-immunotherapy with nivolumab or pembrolizumab regardless of their BRAF status (melanoma)

Exclusion Criteria:

* Segmental or mixed vitiligo (vitiligo)
* Photodermatosis or taking a photosensitizing treatment (vitiligo)
* Patient being allergic to gluten (vitiligo)
* Melanoma of unknown origin (melanoma)
* Ocular melanoma or mucous melanoma (melanoma)
* Patient with brain metastases, symptomatic or not (melanoma)
* Disease not measurable according to RECIST 1.1 criteria (melanoma)
* Patient for whom a combination of anti-PD1 and anti-CTLA-4 immunotherapy is being considered. (melanoma)
* Active autoimmune disease: chronic inflammatory bowel disease and patients with autoimmune disease that is or has been symptomatic
* Patients with autoimmune motor neuropathy
* Concomitant intake of oral immunosuppressive therapy or topical corticosteroid therapy (on vitiligo lesions) or systemic
* Organ transplant patients (kidney, liver, lung, heart, etc.)
* Patient with a history of clinically significant allergy
* History of treatment with anti-CTLA-4, anti-PD-1 or anti-PD-L1, including in an adjuvant situation
* HIV and / or HCV and / or HBV positive serologies
* Patient's refusal to do an HIV, HBV, HCV serology
* Vulnerable people (minors, patients under guardianship or guardianship, deprived of their liberty, under the protection of justice, etc.)
* Patient participating or having participated in another clinical drug trial during the month preceding inclusion
* Women who are pregnant or breastfeeding or who planned to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Changes in blood ITGBL1 expression during immunotherpay | 12 months
  ITGBL1 expression will be measured from the plasma of patients and compared immunotherpy response based on scanner analysis according to RECIST1.1 criteria, and compared to ITGBL1 expression in vitiligo patients or healthy controls

SECONDARY OUTCOMES:
Changes in cytokine CXCL9 expression in plasma | 12 months
  Elisa of different cytokines will be assessed in ng/ml from plasma of patients with melanoma, vitiligo or healthy controls
Changes in cytokine CXCL10 expression in plasma | 12 months
  Elisa of different cytokines will be assessed in ng/ml from plasma of patients with melanoma, vitiligo or healthy controls
Immune cells activity | 12 months
  Immune cells will be isolated from the blood of all subjects and lytic activity against tumor cells will be assessed and compared to immune system activity response from the same patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region, France

IPD SHARING:
Plan to Share IPD: No